CLINICAL TRIAL: NCT01860950
Title: Effects of Transcranial Direct Current Stimulation on Pain Perception
Acronym: tDCS-CBT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: Pro00019694
Record Dates: First submitted 2013-05-21; First posted 2013-05-23 (Estimated); Results first posted 2018-12-04 (Actual); Last update posted 2018-12-04 (Actual); Status verified 2018-12

CONDITIONS: Pain
Keywords: Healthy Adults; Pain Perception
MeSH Terms: conditions — Pain | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- anodal tDCS plus BCI (Active Comparator): Participants underwent Brief Cognitive intervention (BCI) during a single 20-minute session of transcranial direct current stimulation (tDCS) with the anode electrode placed over the left DLPFC and the cathode electrode attached to the right shoulder (Brand Phoresor-II Auto) . BCI entails listening to a 3-minute audio recording designed to mimic key components of cognitive behavioral therapy (CBT) for pain.
  Interventions: Device: anodal tDCS
- anodal tDCS plus pain-education (Active Comparator): Participants were provided pain education during a single 20-minute session of transcranial direct current stimulation (tDCS) with the anode electrode placed over the left DLPFC and the cathode electrode attached to the right shoulder.
  Pain Education information included Pain Physiology, info on the Gate Theory of Pain, and Central Pain Processing.
  Interventions: Device: anodal tDCS
- cathodal tDCS plus BCI (Experimental): Participants underwent Brief Cognitive intervention (BCI) during a single 20-minute session of transcranial direct current stimulation (tDCS) with the anode attached to the right shoulder and the cathode electrode placed over the left DLPFC. BCI entails listening to a 3-minute audio recording designed to mimic key components of cognitive behavioral therapy (CBT) for pain.
  Interventions: Device: cathodal tDCS
- cathodal tDCS plus pain-education (Experimental): Participants were provided pain education during a single 20-minute session of transcranial direct current stimulation (tDCS) with the anode electrode attached to the right shoulder and the cathode electrode was placed over the left DLPFC. Pain Education information included Pain Physiology, info on the Gate Theory of Pain, and Central Pain Processing.
  Interventions: Device: cathodal tDCS
- sham tDCS plus BCI (Sham Comparator): Participants underwent Brief Cognitive intervention (BCI) during 20 minutes of sham tDCS. For sham, the device was turned on for 30 seconds to temporarily mimic tingling and skin sensations of real tDCS and then ramped-down to 0mA for the duration of the 20-minute session.
  Interventions: Device: sham tDCS
- sham tDCS plus pain-education (Sham Comparator): Participants were provided pain education during 20 minutes of sham tDCS. For sham, the device was turned on for 30 seconds to temporarily mimic tingling and skin sensations of real tDCS and then ramped-down to 0mA for the duration of the 20-minute session. Pain Education information included Pain Physiology, info on the Gate Theory of Pain, and Central Pain Processing.
  Interventions: Device: sham tDCS

INTERVENTIONS:
Device: anodal tDCS — a single 20-minute session of transcranial direct current stimulation (tDCS) with the anode electrode placed over the left DLPFC and the cathode electrode attached to the right shoulder
  Other Names: Transcranial Direct Current Stimulation; Phoresor-II Auto
  Arms: anodal tDCS plus BCI; anodal tDCS plus pain-education
Device: cathodal tDCS — a single 20-minute session of transcranial direct current stimulation (tDCS) with the anode attached to the right shoulder and the cathode electrode placed over the left DLPFC.
  Other Names: Transcranial Direct Current Stimulation; Phoresor-II Auto
  Arms: cathodal tDCS plus BCI; cathodal tDCS plus pain-education
Device: sham tDCS — Participants were provided pain education during 20 minutes of sham tDCS. For sham, the device was turned on for 30 seconds to temporarily mimic tingling and skin sensations of real tDCS and then ramped-down to 0mA for the duration of the 20-minute session
  Other Names: Transcranial Direct Current Stimulation; Phoresor-II Auto
  Arms: sham tDCS plus BCI; sham tDCS plus pain-education

SUMMARY:
The purpose of this study is to determine whether a new medical technology can temporarily alter pain perception. The new technology is called Transcranial direct current stimulation (tDCS).

DETAILED DESCRIPTION:
Healthy subjects underwent thermal pain tolerance testing pre- and post intervention. The intervention includes either anodal, cathodal, or sham tDCS for 20 minutes during a pain cognitive intervention [either brief cognitive intervention (BCI) or general pain education]. The tDCS brand was the Phoresor-II Auto (Model PM850, Iomed, Salt Lake City Utah, USA) and the current was set to 2.0mA. Electrodes were 4x4 cm sponge electrodes soaked in sterile saline. For anodal and cathodal tDCS, One electrode was placed over the left DLPFC (F3 from the EEG 10-20 system) located via the Beam F3 measurement system and the other electrode was attached to the right shoulder. For sham tDCS, the device was turned on for 30 seconds to temporarily mimic tingling and skin sensations of real tDCS and then ramped-down to 0mA for the duration of the 20-minute session.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria:

* 100 Health Individuals recruited from Charleston ,SC

Exclusion Criteria:

* Can not be pregnant
* No history of Depression, chronic pain, Seizers, suicidal implanted metal devices, history of brain surgery, loss of consciousness.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Borckardt, Ph.D., Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Anodal tDCS Plus BCI: Participants underwent Brief Cognitive intervention (BCI) during a single 20-minute session of transcranial direct current stimulation (tDCS) with the anode electrode placed over the left DLPFC and the cathode electrode attached to the right shoulder. BCI entails listening to a 3-minute audio recording designed to mimic key components of cognitive behavioral therapy (CBT) for pain.
  anodal tDCS: a single 20-minute session of transcranial direct current stimulation (tDCS) with the anode electrode placed over the left DLPFC and the cathode electrode attached to the right shoulder
- Anodal tDCS Plus Pain-education: Participants were provided pain education during a single 20-minute session of transcranial direct current stimulation (tDCS) with the anode electrode placed over the left DLPFC and the cathode electrode attached to the right shoulder.
  Pain Education information included Pain Physiology, info on the Gate Theory of Pain, and Central Pain Processing.
  anodal tDCS: a single 20-minute session of transcranial direct current stimulation (tDCS) with the anode electrode placed over the left DLPFC and the cathode electrode attached to the right shoulder
Period: Overall Study
Arm/Group | Anodal tDCS Plus BCI | Anodal tDCS Plus Pain-education | Cathodal tDCS Plus BCI | Cathodal tDCS Plus Pain-education | Sham tDCS Plus BCI | Sham tDCS Plus Pain-education
Started | 14 | 15 | 10 | 13 | 14 | 13
Completed | 14 | 15 | 10 | 13 | 14 | 13
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Anodal tDCS Plus BCI | Anodal tDCS Plus Pain-education | Cathodal tDCS Plus BCI | Cathodal tDCS Plus Pain-education | Sham tDCS Plus BCI | Sham tDCS Plus Pain-education | Total
Number analyzed (Participants) | 14 | 15 | 10 | 13 | 14 | 13 | 79
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 14 | 15 | 10 | 13 | 14 | 13 | 79
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.43 (9.27) | 32.60 (11.59) | 27.80 (6.89) | 28.46 (7.24) | 29.93 (8.82) | 38.85 (12.49) | 35 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 6 | 8 | 10 | 10 | 53
  Male | 5 | 5 | 4 | 5 | 4 | 3 | 26
Region of Enrollment [Number; unit: participants]
  United States | 14 | 15 | 10 | 13 | 14 | 13 | 79

OUTCOME MEASURES:

1. Primary Outcome: Pre-Intervention Pain Tolerance
Description: Participants will undergo comprehensive laboratory pain assessment including hot and cold, sensory and pain threshold assessment using the Method of Limits with the Pathway Thermo-sensory Analyzer System (Medoc Inc., NC) which is specifically designed for assessing laboratory pain perception.
Time Frame: Duration of the study visit, approximately 2 hours
Measure: Mean (Standard Deviation); unit: celcius
Arm/Group | Anodal tDCS Plus BCI | Anodal tDCS Plus Pain-education | Cathodal tDCS Plus BCI | Cathodal tDCS Plus Pain-education | Sham tDCS Plus BCI | Sham tDCS Plus Pain-education
Number analyzed (Participants) | 14 | 15 | 10 | 13 | 14 | 13
celcius | 46.49 (1.51) | 47.06 (0.92) | 46.16 (2.15) | 46.82 (2.19) | 46.66 (1.36) | 47.33 (1.04)

2. Primary Outcome: Post-Intervention Pain Tolerance
Description: as for outcome 1
Time Frame: Duration of the study visit, approximately 2 hours
Measure: Mean (Standard Deviation); unit: celcius
Arm/Group | Anodal tDCS Plus BCI | Anodal tDCS Plus Pain-education | Cathodal tDCS Plus BCI | Cathodal tDCS Plus Pain-education | Sham tDCS Plus BCI | Sham tDCS Plus Pain-education
Number analyzed (Participants) | 14 | 15 | 10 | 13 | 14 | 13
celcius | 47.52 (0.98) | 47.11 (1.07) | 47.53 (1.85) | 47.72 (1.72) | 47.47 (1.39) | 47.27 (0.88)

3. Secondary Outcome: Percentage of Participants That Correctly Guessed Condition Assignment
Description: Participants guessed whether they received real tDCS or Sham tDCS. The base-rate for correctly guessing real versus sham was 50%.
Time Frame: 2 hours
Measure: Number; unit: percentage of participants
Groups:
- All Participants: At the end of the laboratory session, participants were asked to indicate whether they thought they received real or sham tDCS. The base-rate for correctly guessing real versus sham was 50%.
Arm/Group | All Participants
Number analyzed (Participants) | 79
percentage of participants | 56

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Anodal tDCS Plus BCI | Anodal tDCS Plus Pain-education | Cathodal tDCS Plus BCI | Cathodal tDCS Plus Pain-education | Sham tDCS Plus BCI | Sham tDCS Plus Pain-education
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/15 | 0/10 | 0/13 | 0/14 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/15 | 0/10 | 0/13 | 0/14 | 0/13
Other Adverse Events (participants affected / at risk) | 0/14 | 0/15 | 0/10 | 0/13 | 0/14 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-07-18): https://cdn.clinicaltrials.gov/large-docs/50/NCT01860950/Prot_SAP_000.pdf
  • Informed Consent Form (2016-08-02): https://cdn.clinicaltrials.gov/large-docs/50/NCT01860950/ICF_001.pdf